CLINICAL TRIAL: NCT03640052
Title: Pharmacological Activation of Hypoglossal Motor Nucleus for Obstructive Sleep Apnea
Brief Title: Pharmacological Activation of HMN for OSA
Acronym: OSA12
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Luigi Taranto Montemurro, Principal investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001201
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo capsule 1 time before bedtime
  Interventions: Drug: Placebo oral capsule
- LTM1201L (Active Comparator): LTM1201L capsule 1 time before bedtime
  Interventions: Drug: LTM1201L
- LTM1201LN (Active Comparator): LTM1201LN capsule 1 time before bedtime
  Interventions: Drug: LTM1201LN
- LTM1201LB (Active Comparator): LTM1201LB capsule 1 time before bedtime
  Interventions: Drug: LTM1201LB
- LTM1201LD (Active Comparator): LTM1201LD capsule 1 time before bedtime
  Interventions: Drug: LTM1201LD

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo capsule before sleep
  Arms: Placebo
Drug: LTM1201L — LTM1201L capsule before sleep
  Arms: LTM1201L
Drug: LTM1201LN — LTM1201LN capsule before sleep
  Arms: LTM1201LN
Drug: LTM1201LB — LTM1201LB capsule before sleep
  Arms: LTM1201LB
Drug: LTM1201LD — LTM1201LD capsule before sleep
  Arms: LTM1201LD

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal subjects. In this protocol the investigators will test the effect of LTM1201L, LTM1201LN, LTM1201LB, LTM1201LD administered before sleep on OSA phenotype traits and OSA severity during sleep.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 10 events/h during NREM supine sleep

Exclusion Criteria:

* Any medical condition other than well controlled hypertension and mild diabetes.
* Any medication known to influence breathing, sleep/arousal, or muscle physiology.
* Claustrophobia.
* Inability to sleep supine.
* Allergy to any of the medications tested in the protocol.
* History of kidney stones, hypercalcemia, primary hyperparathyroidism, sarcoidosis, hypervitaminosis D.
* Individuals with underlying cardiac disease, such as arrhythmias.
* Individuals taking psychiatric medications, such as an MAO-I, SSRI or SNRI, or any of the studied medications for medical care.
* For women: Pregnancy.
* Pulmonary hypertension
* Severe OSA with a mean SaO2 lower than 88%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First: Placebo administered before sleep for 1 night, followed by LTM1201L, LTM1201LD, LTM1201LN and LTM1201LB, administered 1 week apart in the hospital
- LTM1201L First: LTM1201L administered before sleep for 1 night, followed by LTM1201LD, LTM1201LN, LTM1201LB and Placebo, administered 1 week apart in the hospital
- LTM1201LD First: LTM1201LD administered before sleep for 1 night, followed by LTM1201LN, LTM1201LB, Placebo and LTM1201L, administered 1 week apart in the hospital
- LTM1201LN First: LTM1201LN administered before sleep for 1 night, followed by LTM1201LB, Placebo, LTM1201L and LTM1201LD administered 1 week apart in the hospital
- LTM1201LB First: LTM1201LB administered before sleep for 1 night, followed by Placebo, LTM1201L, LTM1201LD and LTM1201LN administered 1 week apart in the hospital
Period: Overall Study
Arm/Group | Placebo First | LTM1201L First | LTM1201LD First | LTM1201LN First | LTM1201LB First
Started | 2 | 1 | 1 | 1 | 1
Completed | 2 | 0 (the patient performed 4 out of 5 nights) | 1 | 1 | 1
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.5 [47 to 54.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI, Average Number of Events for Every Hour of Sleep)
Description: Based on previous studies the investigators anticipate that active comparators will reduce AHI more effectively in subjects with moderate sleep apnea and low-to-moderate collapsibility (Vpassive >50% of eupneic values). Higher AHI indicates more severe OSA, usually ranging between 10 to 110 events/hour.
Time Frame: 1 night
Measure: Mean (Standard Error); unit: events/hour of sleep
Arm/Group | Placebo | LTM1201L | LTM1201LN | LTM1201LB | LTM1201LD
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
events/hour of sleep | 20.8 (8) | 24.4 (11.3) | 18.8 (11.3) | 14 (11.3) | 9.1 (11.9)
Statistical Analysis 1: Comparison: LTM1201L; mean difference vs Placebo; Test type: Superiority; p > 0.5, Mixed Models Analysis; Mean Difference (Final Values) = 3.6
Statistical Analysis 2: Comparison: LTM1201LN; mean difference vs Placebo; Test type: Superiority; p > 0.5, Mixed Models Analysis; Mean Difference (Net) = -2
Statistical Analysis 3: Comparison: LTM1201LB; mean difference vs Placebo; Test type: Superiority; p > 0.5, Mixed Models Analysis; Mean Difference (Net) = -6.8
Statistical Analysis 4: Comparison: LTM1201LD; mean difference vs Placebo; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Net) = -11.7

2. Secondary Outcome: Collapsibility of the Upper Airway: VActive (L/Min)
Description: VActive: ventilation when ventilatory drive is high and pharyngeal dilator muscles are relatively active.
Time Frame: 1 night
Measure: Mean (Standard Error); unit: Liters/minute
Arm/Group | Placebo | LTM1201L | LTM1201LN | LTM1201LB | LTM1201LD
Number analyzed (Participants) | 6 | 5 | 6 | 3 | 6
Liters/minute | 2.657 (0.6865) | 3.856 (1.04) | 3.822 (1.049) | 6.008 (1.11) | 3.091 (1.161)
Statistical Analysis 1: Comparison: Placebo vs LTM1201L vs LTM1201LN vs LTM1201LB vs LTM1201LD; Test type: Superiority; p = 0.12, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 night
Arm/Group | Placebo | LTM1201L | LTM1201LN | LTM1201LB | LTM1201LD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 5/6 | 3/5 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | LTM1201L (N=6) | LTM1201LN (N=6) | LTM1201LB (N=5) | LTM1201LD (N=6)
Dry mouth (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 3 (3) — Dry mouth
insomnia (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT03640052/Prot_SAP_000.pdf